CLINICAL TRIAL: NCT02389400
Title: Efficacy and Tolerance of Combination Chemotherapy With Methotrexate and Cytosine Arabinoside in Newly Diagnosed Adult With Langerhans Cell Histiocytosis
Brief Title: Methotrexate and Cytosine in Adult Langerhans Cell Histiocytosis
Acronym: MAALCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALCH-MA-001
Record Dates: First submitted 2015-02-09; First posted 2015-03-17 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2017-08

CONDITIONS: Langerhans Cell Histiocytosis
Keywords: adult with Langerhans cell histiocytosis; newly diagnosed; methotrexate; cytosine arabinoside
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Methotrexate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental arm (Experimental): methotrexate,1g/m2,iv.d1 cytosine arabinoside,0.1g/m2,iv.,d1-5
  Interventions: Drug: methotrexate

INTERVENTIONS:
Drug: methotrexate — Single Group Assignment
  Other Names: cytosine arabinoside

SUMMARY:
Study Type: Interventional

Study Design:

Endpoint Classification: Efficacy Study Intervention Model: Single Group Assignment Masking: Open Label Primary Purpose: Treatment purpose: This single arm clinical trial is studying efficacy and tolerance of combination chemotherapy with methotrexate and cytosine arabinoside in newly diagnosed adult with Langerhans cell histiocytosis.

DETAILED DESCRIPTION:
This single arm clinical trial is studying efficacy and tolerance of combination chemotherapy with methotrexate and cytosine arabinoside in newly diagnosed adult with Langerhans cell histiocytosis.

ELIGIBILITY:
Inclusion Criteria:

1.DISEASE CHARACTERISTICS:

* Histopathologically confirmed diagnosis of Langerhans cell histiocytosis according to the criteria defined by the Histiocyte Society
* Demonstration of CD1a antigenic determinants on the surface of lesional cells (by immunocytology or immunohistology) or Birbeck granules in lesional cells by electron microscopy
* Considered at risk or low risk according to the following criteria:

  * Multi-system at risk disease, defined as involvement of one or more risk organs (i.e., hematopoietic system, liver, spleen, or lungs)

    1.No single-system lung involvement
  * Multi-system low-risk disease

    1.Multiple organs involved but without involvement of risk organs
  * Single-system disease 1.Multifocal bone disease (i.e., lesions in 2 or more different bones) 2.Localized special site involvement, such as CNS-risk lesions with intracranial soft tissue extension or vertebral lesions with intraspinal soft tissue extension 3.Vault lesions are not regarded as CNS-risk lesions 2.PATIENT CHARACTERISTICS:

    1. Not pregnant or nursing
    2. Negative pregnancy test
    3. Fertile patients must use effective contraception 3.PRIOR CONCURRENT THERAPY:

    <!-- -->

    1. No prior treatment for Langerhans cell histiocytosis

Exclusion Criteria:

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-01; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
disease free survival | 5 years
  time from treatment to disease progression

SECONDARY OUTCOMES:
overall free survival | 5 years
  time from treatment to die

OTHER OUTCOMES:
Response | 2 years
  The bone lesion response and the central nervous system（CNS）lesions response

CONTACTS AND LOCATIONS:
Overall Officials: minghui Duan, Dr., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking union medical college hospital, Beijing, China

REFERENCES:
- [Derived] Han X, Ouyang M, Duan M, Zhang W, Zhu T, Li J, Wang S, Zhou D. The combination of methotrexate and cytosine arabinoside in newly diagnosed adult Langerhans cell histiocytosis: a prospective phase II interventional clinical trial. BMC Cancer. 2020 May 18;20(1):433. doi: 10.1186/s12885-020-06872-8. PMID 32423455